CLINICAL TRIAL: NCT03333590
Title: Phase I/IIa Gene Transfer Clinical Trial for Duchenne Muscular Dystrophy Using rAAVrh74.MCK.GALGT2
Brief Title: Gene Transfer Clinical Trial to Deliver rAAVrh74.MCK.GALGT2 for Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kevin Flanigan (Other)
Responsible Party: Sponsor-Investigator, Kevin Flanigan, Professor of Pediatrics, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GALGT2 Gene Therapy for DMD
Record Dates: First submitted 2017-11-01; First posted 2017-11-07 (Actual); Results first posted 2022-04-25 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD; Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Intervention Model Description: This is a dose escalation trial that will begin with the minimal efficacious dose as determined by preclinical studies and approved by the FDA. During the course of the trial, if safety is shown the dose will be escalated according to the clinical protocol.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Minimal Efficacious Dose) rAAVrh74.MCK.GALGT2 (Experimental): N = 3 [2.5 x E13 vg/kg per leg, delivered bilaterally (total 5.0 x E13 vg/kg)]
  Interventions: Biological: rAAVrh74.MCK.GALGT2
- Cohort 2 (Dose Escalation) rAAVrh74.MCK.GALGT2 (Experimental): N=3 [5 x E13 vg/kg per leg, delivered bilaterally (total 1.0 x E14 vg/kg)]
  Interventions: Biological: rAAVrh74.MCK.GALGT2

INTERVENTIONS:
Biological: rAAVrh74.MCK.GALGT2 — Adeno-associated virus serotype rh74 carrying the GALGT2 gene under the control of a MCK promoter (rAAVrh74.MCK.GALGT2) will be delivered one time to each of the lower limbs through the femoral artery using an intravascular limb infusion technique (ILI)

SUMMARY:
The proposed clinical trial study of rAAVrh74.MCK.GALGT2 for duchenne muscular dystrophy (DMD) patients. There will be a modified intravascular limb infusion (ILI) procedure that will be used to sequentially deliver vector to each whole lower limb of DMD subjects via a major lower limb artery.

DETAILED DESCRIPTION:
This is an open-label, dose escalation trial where the vector will be delivered via the femoral artery to the muscles of both legs of DMD subjects.

The primary objective of this study is the assessment of the safety of intravascular administration of rAAVrh74.MCK.GALGT2 to DMD patients. Safety endpoints will be assessed by changes in hematology, serum chemistry, urinalysis, immunologic response to rAAVrh74 and GALGT2, and reported history and observations of symptoms. Efficacy measures will be used as secondary outcome for this disorder including a combination of functional 6 minute walk test (6MWT) and direct muscle testing for strength (MVICT) of lower limb muscles.

Subjects will be evaluated at baseline, infusion visit (days 0-2), and return for follow up visits on days 7, 14, 30, 60, 90, and 180 and months 12, 18 and 24

ELIGIBILITY:
Inclusion Criteria

* Ambulant patients age 4 years or older
* Confirmed mutations in the DMD gene using a clinical accepted technique that completely defines the mutation 1,2
* • Measurably impaired muscle function (defined as less than 80% of the predicted value for 100 MWT), but with sufficient muscle preservation to ensure assessment of muscle transfection based on clinical evaluation by the PI and expert colleagues. This degree of preservation will include:

  * Ability to extend the knee fully against gravity
  * Preserved ambulation with ability to walk ≥ 350 meters during the 6MWT
  * A magnetic resonance image of the quadriceps showing preservation of sufficient muscle mass to permit transfection
* Males of any ethnic group will be eligible
* Ability to cooperate with muscle testing
* Stable daily dose of corticosteroid therapy (including either prednisone, prednisolone, deflazacort or their generic forms) for 12 weeks prior to gene transfer

Exclusion Criteria

* Active viral infection based on clinical observations
* The presence of a DMD mutation without weakness or loss of function
* Subject is amenable to or is currently being treated with eteplirsen
* Symptoms or signs of cardiomyopathy, including:

  * Dyspnea on exertion, pedal edema, shortness of breath upon lying flat, or rales at the base of the lungs
  * Echocardiogram with ejection fraction below 40%
* Serological evidence of HIV infection, or Hepatitis B or C infection
* Diagnosis of (or ongoing treatment for) an autoimmune disease
* Persistent leukopenia or leukocytosis (WBC ≤ 3.5 K/µL or ≥ 20.0 K/µL) or an absolute neutrophil count < 1.5K/µL
* Concomitant illness or requirement for chronic drug treatment that in the opinion of the PI creates unnecessary risks for gene transfer
* Subjects with rAAVrh74 binding antibody titers ≥ 1:50 as determined by ELISA immunoassay
* Presence of circulating anti-Sda antibodies as determined by study approved laboratory
* Abnormal laboratory values in the clinically significant range, based upon normal values in the Nationwide Children's Hospital Laboratory

Min Age: 4 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Flanigan, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Chicoine LG, Rodino-Klapac LR, Shao G, Xu R, Bremer WG, Camboni M, Golden B, Montgomery CL, Shontz K, Heller KN, Griffin DA, Lewis S, Coley BD, Walker CM, Clark KR, Sahenk Z, Mendell JR, Martin PT. Vascular delivery of rAAVrh74.MCK.GALGT2 to the gastrocnemius muscle of the rhesus macaque stimulates the expression of dystrophin and laminin alpha2 surrogates. Mol Ther. 2014 Apr;22(4):713-24. doi: 10.1038/mt.2013.246. Epub 2013 Oct 22. PMID 24145553
- [Background] Flanigan KM, Dunn DM, von Niederhausern A, Soltanzadeh P, Gappmaier E, Howard MT, Sampson JB, Mendell JR, Wall C, King WM, Pestronk A, Florence JM, Connolly AM, Mathews KD, Stephan CM, Laubenthal KS, Wong BL, Morehart PJ, Meyer A, Finkel RS, Bonnemann CG, Medne L, Day JW, Dalton JC, Margolis MK, Hinton VJ; United Dystrophinopathy Project Consortium; Weiss RB. Mutational spectrum of DMD mutations in dystrophinopathy patients: application of modern diagnostic techniques to a large cohort. Hum Mutat. 2009 Dec;30(12):1657-66. doi: 10.1002/humu.21114. PMID 19937601
- [Background] Flanigan KM, von Niederhausern A, Dunn DM, Alder J, Mendell JR, Weiss RB. Rapid direct sequence analysis of the dystrophin gene. Am J Hum Genet. 2003 Apr;72(4):931-9. doi: 10.1086/374176. Epub 2003 Mar 11. PMID 12632325
- [Background] Seinen JM, Hoekstra HJ. Isolated limb perfusion of soft tissue sarcomas: a comprehensive review of literature. Cancer Treat Rev. 2013 Oct;39(6):569-77. doi: 10.1016/j.ctrv.2012.10.005. Epub 2012 Dec 8. PMID 23232098
- [Background] Rodino-Klapac LR, Janssen PM, Montgomery CL, Coley BD, Chicoine LG, Clark KR, Mendell JR. A translational approach for limb vascular delivery of the micro-dystrophin gene without high volume or high pressure for treatment of Duchenne muscular dystrophy. J Transl Med. 2007 Sep 24;5:45. doi: 10.1186/1479-5876-5-45. PMID 17892583
- [Background] Rodino-Klapac LR, Montgomery CL, Bremer WG, Shontz KM, Malik V, Davis N, Sprinkle S, Campbell KJ, Sahenk Z, Clark KR, Walker CM, Mendell JR, Chicoine LG. Persistent expression of FLAG-tagged micro dystrophin in nonhuman primates following intramuscular and vascular delivery. Mol Ther. 2010 Jan;18(1):109-17. doi: 10.1038/mt.2009.254. Epub 2009 Nov 10. PMID 19904237
- [Background] Rodino-Klapac LR, Montgomery CL, Mendell JR, Chicoine LG. AAV-mediated gene therapy to the isolated limb in rhesus macaques. Methods Mol Biol. 2011;709:287-98. doi: 10.1007/978-1-61737-982-6_19. PMID 21194036
- [Background] Mendell JR, Shilling C, Leslie ND, Flanigan KM, al-Dahhak R, Gastier-Foster J, Kneile K, Dunn DM, Duval B, Aoyagi A, Hamil C, Mahmoud M, Roush K, Bird L, Rankin C, Lilly H, Street N, Chandrasekar R, Weiss RB. Evidence-based path to newborn screening for Duchenne muscular dystrophy. Ann Neurol. 2012 Mar;71(3):304-13. doi: 10.1002/ana.23528. PMID 22451200
- [Background] Brooke MH, Fenichel GM, Griggs RC, Mendell JR, Moxley R, Miller JP, Province MA. Clinical investigation in Duchenne dystrophy: 2. Determination of the "power" of therapeutic trials based on the natural history. Muscle Nerve. 1983 Feb;6(2):91-103. doi: 10.1002/mus.880060204. PMID 6343858
- [Background] Eagle M, Baudouin SV, Chandler C, Giddings DR, Bullock R, Bushby K. Survival in Duchenne muscular dystrophy: improvements in life expectancy since 1967 and the impact of home nocturnal ventilation. Neuromuscul Disord. 2002 Dec;12(10):926-9. doi: 10.1016/s0960-8966(02)00140-2. PMID 12467747
- [Background] Koenig M, Hoffman EP, Bertelson CJ, Monaco AP, Feener C, Kunkel LM. Complete cloning of the Duchenne muscular dystrophy (DMD) cDNA and preliminary genomic organization of the DMD gene in normal and affected individuals. Cell. 1987 Jul 31;50(3):509-17. doi: 10.1016/0092-8674(87)90504-6. PMID 3607877
- [Background] Bonilla E, Samitt CE, Miranda AF, Hays AP, Salviati G, DiMauro S, Kunkel LM, Hoffman EP, Rowland LP. Duchenne muscular dystrophy: deficiency of dystrophin at the muscle cell surface. Cell. 1988 Aug 12;54(4):447-52. doi: 10.1016/0092-8674(88)90065-7. PMID 3042151
- [Background] Oudet C, Hanauer A, Clemens P, Caskey T, Mandel JL. Two hot spots of recombination in the DMD gene correlate with the deletion prone regions. Hum Mol Genet. 1992 Nov;1(8):599-603. doi: 10.1093/hmg/1.8.599. PMID 1363782
- [Background] Beggs AH, Koenig M, Boyce FM, Kunkel LM. Detection of 98% of DMD/BMD gene deletions by polymerase chain reaction. Hum Genet. 1990 Nov;86(1):45-8. doi: 10.1007/BF00205170. PMID 2253937
- [Background] Chamberlain JS, Gibbs RA, Ranier JE, Nguyen PN, Caskey CT. Deletion screening of the Duchenne muscular dystrophy locus via multiplex DNA amplification. Nucleic Acids Res. 1988 Dec 9;16(23):11141-56. doi: 10.1093/nar/16.23.11141. PMID 3205741
- [Background] Lalic T, Vossen RH, Coffa J, Schouten JP, Guc-Scekic M, Radivojevic D, Djurisic M, Breuning MH, White SJ, den Dunnen JT. Deletion and duplication screening in the DMD gene using MLPA. Eur J Hum Genet. 2005 Nov;13(11):1231-4. doi: 10.1038/sj.ejhg.5201465. PMID 16030524
- [Background] Dent KM, Dunn DM, von Niederhausern AC, Aoyagi AT, Kerr L, Bromberg MB, Hart KJ, Tuohy T, White S, den Dunnen JT, Weiss RB, Flanigan KM. Improved molecular diagnosis of dystrophinopathies in an unselected clinical cohort. Am J Med Genet A. 2005 Apr 30;134(3):295-8. doi: 10.1002/ajmg.a.30617. PMID 15723292
- [Background] Mendell JR, Moxley RT, Griggs RC, Brooke MH, Fenichel GM, Miller JP, King W, Signore L, Pandya S, Florence J, et al. Randomized, double-blind six-month trial of prednisone in Duchenne's muscular dystrophy. N Engl J Med. 1989 Jun 15;320(24):1592-7. doi: 10.1056/NEJM198906153202405. PMID 2657428
- [Background] Balaban B, Matthews DJ, Clayton GH, Carry T. Corticosteroid treatment and functional improvement in Duchenne muscular dystrophy: long-term effect. Am J Phys Med Rehabil. 2005 Nov;84(11):843-50. doi: 10.1097/01.phm.0000184156.98671.d0. PMID 16244521
- [Background] Griggs RC, Moxley RT 3rd, Mendell JR, Fenichel GM, Brooke MH, Pestronk A, Miller JP. Prednisone in Duchenne dystrophy. A randomized, controlled trial defining the time course and dose response. Clinical Investigation of Duchenne Dystrophy Group. Arch Neurol. 1991 Apr;48(4):383-8. doi: 10.1001/archneur.1991.00530160047012. PMID 2012511
- [Background] Biggar WD, Harris VA, Eliasoph L, Alman B. Long-term benefits of deflazacort treatment for boys with Duchenne muscular dystrophy in their second decade. Neuromuscul Disord. 2006 Apr;16(4):249-55. doi: 10.1016/j.nmd.2006.01.010. Epub 2006 Mar 20. PMID 16545568
- [Background] Mendell JR, Goemans N, Lowes LP, Alfano LN, Berry K, Shao J, Kaye EM, Mercuri E; Eteplirsen Study Group and Telethon Foundation DMD Italian Network. Longitudinal effect of eteplirsen versus historical control on ambulation in Duchenne muscular dystrophy. Ann Neurol. 2016 Feb;79(2):257-71. doi: 10.1002/ana.24555. Epub 2016 Jan 8. PMID 26573217
- [Background] Mendell JR, Rodino-Klapac LR, Sahenk Z, Roush K, Bird L, Lowes LP, Alfano L, Gomez AM, Lewis S, Kota J, Malik V, Shontz K, Walker CM, Flanigan KM, Corridore M, Kean JR, Allen HD, Shilling C, Melia KR, Sazani P, Saoud JB, Kaye EM; Eteplirsen Study Group. Eteplirsen for the treatment of Duchenne muscular dystrophy. Ann Neurol. 2013 Nov;74(5):637-47. doi: 10.1002/ana.23982. Epub 2013 Sep 10. PMID 23907995
- [Background] Bushby K, Finkel R, Wong B, Barohn R, Campbell C, Comi GP, Connolly AM, Day JW, Flanigan KM, Goemans N, Jones KJ, Mercuri E, Quinlivan R, Renfroe JB, Russman B, Ryan MM, Tulinius M, Voit T, Moore SA, Lee Sweeney H, Abresch RT, Coleman KL, Eagle M, Florence J, Gappmaier E, Glanzman AM, Henricson E, Barth J, Elfring GL, Reha A, Spiegel RJ, O'donnell MW, Peltz SW, Mcdonald CM; PTC124-GD-007-DMD STUDY GROUP. Ataluren treatment of patients with nonsense mutation dystrophinopathy. Muscle Nerve. 2014 Oct;50(4):477-87. doi: 10.1002/mus.24332. PMID 25042182
- [Background] Finkel RS, Flanigan KM, Wong B, Bonnemann C, Sampson J, Sweeney HL, Reha A, Northcutt VJ, Elfring G, Barth J, Peltz SW. Phase 2a study of ataluren-mediated dystrophin production in patients with nonsense mutation Duchenne muscular dystrophy. PLoS One. 2013 Dec 11;8(12):e81302. doi: 10.1371/journal.pone.0081302. eCollection 2013. PMID 24349052
- [Background] Mendell JR, Rodino-Klapac LR, Rosales XQ, Coley BD, Galloway G, Lewis S, Malik V, Shilling C, Byrne BJ, Conlon T, Campbell KJ, Bremer WG, Taylor LE, Flanigan KM, Gastier-Foster JM, Astbury C, Kota J, Sahenk Z, Walker CM, Clark KR. Sustained alpha-sarcoglycan gene expression after gene transfer in limb-girdle muscular dystrophy, type 2D. Ann Neurol. 2010 Nov;68(5):629-38. doi: 10.1002/ana.22251. PMID 21031578
- [Background] Harper SQ, Hauser MA, DelloRusso C, Duan D, Crawford RW, Phelps SF, Harper HA, Robinson AS, Engelhardt JF, Brooks SV, Chamberlain JS. Modular flexibility of dystrophin: implications for gene therapy of Duchenne muscular dystrophy. Nat Med. 2002 Mar;8(3):253-61. doi: 10.1038/nm0302-253. PMID 11875496
- [Background] Gregorevic P, Blankinship MJ, Allen JM, Crawford RW, Meuse L, Miller DG, Russell DW, Chamberlain JS. Systemic delivery of genes to striated muscles using adeno-associated viral vectors. Nat Med. 2004 Aug;10(8):828-34. doi: 10.1038/nm1085. Epub 2004 Jul 25. PMID 15273747
- [Background] Xu R, DeVries S, Camboni M, Martin PT. Overexpression of Galgt2 reduces dystrophic pathology in the skeletal muscles of alpha sarcoglycan-deficient mice. Am J Pathol. 2009 Jul;175(1):235-47. doi: 10.2353/ajpath.2009.080967. Epub 2009 Jun 4. PMID 19498002
- [Background] Xu R, Chandrasekharan K, Yoon JH, Camboni M, Martin PT. Overexpression of the cytotoxic T cell (CT) carbohydrate inhibits muscular dystrophy in the dyW mouse model of congenital muscular dystrophy 1A. Am J Pathol. 2007 Jul;171(1):181-99. doi: 10.2353/ajpath.2007.060927. PMID 17591965
- [Background] Liu G, McNicol PL, Macall P, Bellomo R, Przybylowski G, Bowkett J, Connellan J, McInnes F, Thurlow PJ. The Effect of Preoperative Aspirin and/or Heparin Therapy on Coagulation and Postoperative Blood Loss after Coronary Artery Bypass Surgery. Crit Care Resusc. 1999 Jun;1(2):139. PMID 16602995
- [Background] Veikutiene A, Sirvinskas E, Grybauskas P, Cimbolaityte J, Mongirdiene A, Veikutis V. [Influence of preoperative treatment with aspirin or heparin on platelet function and intensity of postoperative bleeding in early period after coronary artery bypass surgery]. Medicina (Kaunas). 2005;41(7):577-83. Lithuanian. PMID 16062025
- [Background] Sun JC, Crowther MA, Warkentin TE, Lamy A, Teoh KH. Should aspirin be discontinued before coronary artery bypass surgery? Circulation. 2005 Aug 16;112(7):e85-90. doi: 10.1161/CIRCULATIONAHA.105.546697. No abstract available. PMID 16103244
- [Background] Taylor LE, Kaminoh YJ, Rodesch CK, Flanigan KM. Quantification of dystrophin immunofluorescence in dystrophinopathy muscle specimens. Neuropathol Appl Neurobiol. 2012 Oct;38(6):591-601. doi: 10.1111/j.1365-2990.2012.01250.x. PMID 22243335
- [Background] Anthony K, Arechavala-Gomeza V, Taylor LE, Vulin A, Kaminoh Y, Torelli S, Feng L, Janghra N, Bonne G, Beuvin M, Barresi R, Henderson M, Laval S, Lourbakos A, Campion G, Straub V, Voit T, Sewry CA, Morgan JE, Flanigan KM, Muntoni F. Dystrophin quantification: Biological and translational research implications. Neurology. 2014 Nov 25;83(22):2062-9. doi: 10.1212/WNL.0000000000001025. Epub 2014 Oct 29. PMID 25355828

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 2 (Minimal Efficacious Dose) rAAVrh74.MCK.GALGT2: N = 3 [5 x E13 vg/kg per leg, delivered bilaterally (total 1.0 x E14 vg/kg)]
  rAAVrh74.MCK.GALGT2: Adeno-associated virus serotype rh74 carrying the GALGT2 gene under the control of a MCK promoter (rAAVrh74.MCK.GALGT2) will be delivered one time to each of the lower limbs through the femoral artery using an intravascular limb infusion technique (ILI)
Period: Overall Study
Arm/Group | Cohort 1 (Minimal Efficacious Dose) rAAVrh74.MCK.GALGT2 | Cohort 2 (Minimal Efficacious Dose) rAAVrh74.MCK.GALGT2
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: There was not enough clinical vector to dose additional participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Minimal Efficacious Dose) rAAVrh74.MCK.GALGT2 | Cohort 2 (Dose Escalation) rAAVrh74.MCK.GALGT2 | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 9 | 7 | 8 [7 to 9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Unanticipated Grade III or Higher Treatment-Related Toxicities
Time Frame: 2 years
Measure: Number; unit: events
Groups:
- Cohort 1 (Minimal Efficacious Dose): N = 1 [2.5 x E13 vg/kg per leg, delivered bilaterally (total 5.0 x E13 vg/kg)]
  rAAVrh74.MCK.GALGT2: Adeno-associated virus serotype rh74 carrying the GALGT2 gene under the control of a MCK promoter (rAAVrh74.MCK.GALGT2) will be delivered one time to each of the lower limbs through the femoral artery using an intravascular limb infusion technique (ILI)
- Cohort 2: N = 1 [5 x E13 vg/kg per leg, delivered bilaterally (total 1.0 x E14 vg/kg)]
  rAAVrh74.MCK.GALGT2: Adeno-associated virus serotype rh74 carrying the GALGT2 gene under the control of a MCK promoter (rAAVrh74.MCK.GALGT2) will be delivered one time to each of the lower limbs through the femoral artery using an intravascular limb infusion technique (ILI)
Arm/Group | Cohort 1 (Minimal Efficacious Dose) | Cohort 2
Number analyzed (Participants) | 1 | 1
events | 0 | 0

2. Secondary Outcome: Expression of GALGT2 as Demonstrated by Immunofluorescent Staining With Anti-CT Epitope Antibodies or WFA Lectin in Muscle Biopsy Sections at 120 Days Post Injection (Cohort 1) and 90 Days Post-injection (Cohort 2).
Description: Percentage of fibers expressing GALGT2 in each biopsy sample.
Time Frame: Day 90 (Cohort 2) and Day 120 (Cohort 1)
Measure: Number; unit: Percentage of Positive Fibers
Units Other Than Participants: Biopsies
Arm/Group | Cohort 1 (Minimal Efficacious Dose) | Cohort 2
Number analyzed (Participants) | 1 | 1
Number analyzed (Biopsies) | 1 | 1
Percentage of Positive Fibers | 1.95 | 1.72

3. Secondary Outcome: GALGT2 Protein Expression Quantified by Western Blot and Assessed by Densitometry in Muscle Biopsy Tissue at 120 Days Post-injection (Cohort 1) and 90 Days Post-injection (Cohort 2)
Time Frame: Day 90 (Cohort 2) and Day 120 (Cohort 1)
Measure: Number; unit: ng/mg total protein
Units Other Than Participants: Biopsies
Arm/Group | Cohort 1 (Minimal Efficacious Dose) | Cohort 2
Number analyzed (Participants) | 1 | 1
Number analyzed (Biopsies) | 1 | 1
ng/mg total protein | 12 | 14.6

4. Other Pre Specified Outcome: Number of Meters Walked During the 6 Minute Walk Test
Time Frame: Day 90 (Cohort 2) and Day 120 (Cohort 1) and Day 180 for both cohorts
Measure: Number; unit: meters
Groups:
- Cohort 2 (Minimal Efficacious Dose): N = 1 [5 x E13 vg/kg per leg, delivered bilaterally (total 1.0 x E14 vg/kg)]
  rAAVrh74.MCK.GALGT2: Adeno-associated virus serotype rh74 carrying the GALGT2 gene under the control of a MCK promoter (rAAVrh74.MCK.GALGT2) will be delivered one time to each of the lower limbs through the femoral artery using an intravascular limb infusion technique (ILI)
Arm/Group | Cohort 1 (Minimal Efficacious Dose) | Cohort 2 (Minimal Efficacious Dose)
Number analyzed (Participants) | 1 | 1
meters
  Day 90 (Cohort 2) /Day 120 (Cohort 1) | 320 | 405
  Day 180 | 324 | 416

5. Other Pre Specified Outcome: Strength of the Bilateral Knee Flexors and Extensors During the Maximal Voluntary Isometric Strength Test.
Time Frame: Days 90 (Cohort 2), 120 (Cohort 1) and both Cohorts at Day 180, Months 12, 18 and 24
Measure: Number; unit: kg
Arm/Group | Cohort 1 (Minimal Efficacious Dose) | Cohort 2
Number analyzed (Participants) | 1 | 1
kg
  Day 90/Day 120-Right Knee Extension | 7.42 | 7.04
  Day 90/Day 120-Right Knee Flexion | 6.06 | 8.12
  Day 90/Day 120- Left Knee Extension | 8.78 | 5.9
  Day 90/Day 120-Left Knee Flexion | 6.12 | 8.4
  Day 180-Right Knee Extension | 7.13 | 9.73
  Day 180-Right Knee Flexion | 6.1 | 4.24
  Day 180-Left Knee Extension | 8.66 | 8.19
  Day 180-Left Knee Flexion | 6.69 | 5.25
  Month 12-Right Knee Extension | 7.49 | 9.85
  Month 12-Right Knee Flexion | 5.67 | 5.85
  Month 12-Left Knee Extension | 7.5 | 8.02
  Month 12-Left Knee Flexion | 5.32 | 5.12
  Month 18-Right Knee Extension | 4.55 | 7.67
  Month 18-Right Knee Flexion | 6.11 | 6.89
  Month 18-Left Knee Extension | 4.96 | 7.34
  Month 18-Left Knee Flexion | 6.26 | 6.08
  Month 24-Right Knee Extension | 5.06 | 9.81
  Month 24-Right Knee Flexion | 4.41 | 5.04
  Month 24-Left Knee Extension | 6.93 | 5.21
  Month 24-Left Knee Flexion | 4.17 | 4.87

6. Other Pre Specified Outcome: Time Taken to Walk 100 Meters During the 100 Meter Walk Test.
Time Frame: Days 90 (Cohort 2), 120 (Cohort 1); both Cohorts at Day 180, Months 12, 18 and Cohort 2 at Month 24
Population: There is no data for Cohort 1, Month 24 because single subject was unable to perform the test.
Measure: Number; unit: seconds
Groups:
- Cohort 2: rAAVrh74.MCK.GALGT2: Adeno-associated virus serotype rh74 carrying the GALGT2 gene under the control of a MCK promoter (rAAVrh74.MCK.GALGT2) will be delivered one time to each of the lower limbs through the femoral artery using an intravascular limb infusion technique (ILI)
Arm/Group | Cohort 1 (Minimal Efficacious Dose) | Cohort 2
Number analyzed (Participants) | 1 | 1
seconds
  Day 90/Day 120 | 98.2 | 56.1
  Day 180 | 110.9 | 44.9
  Month 12 | 144.5 | 44.7
  Month 18 | 167.8 | 65.6
  Month 24: number analyzed (Participants) | 0 | 1
  Month 24 |  | 48.4

7. Other Pre Specified Outcome: Score of Muscle Function Using the The North Star Ambulatory Assessment (NSAA).
Description: The NSAA provides a score between 0 and 34 where higher numbers represent greater muscle function.
Time Frame: Days 90 (Cohort 2), 120 (Cohort 1) and both Cohorts at Day 180, Months 12, 18 and 24
Measure: Number; unit: score on a scale
Arm/Group | Cohort 1 (Minimal Efficacious Dose) | Cohort 2
Number analyzed (Participants) | 1 | 1
score on a scale
  Day 90/Day 120 | 16 | 21
  Day 180 | 14 | 23
  Month 12 | 10 | 23
  Month 18 | 6 | 23
  Month 24 | 2 | 23

ADVERSE EVENTS:
Time Frame: Adverse events started to be collected on Day 0 as defined by the day of Gene Transfer and continued through during the active 2-year period following gene transfer as described in the protocol.
Groups:
- Cohort 1 (Minimal Efficacious Dose) rAAVrh74.MCK.GALGT2: N = 1 [2.5 x E13 vg/kg per leg, delivered bilaterally (total 5.0 x E13 vg/kg)]
  rAAVrh74.MCK.GALGT2: Adeno-associated virus serotype rh74 carrying the GALGT2 gene under the control of a MCK promoter (rAAVrh74.MCK.GALGT2) will be delivered one time to each of the lower limbs through the femoral artery using an intravascular limb infusion technique (ILI)
- Cohort 1 rAAVrh74.MCK.GALGT2: N = 1 [5 x E13 vg/kg per leg, delivered bilaterally (total 1.0 x E14 vg/kg)]
  rAAVrh74.MCK.GALGT2: Adeno-associated virus serotype rh74 carrying the GALGT2 gene under the control of a MCK promoter (rAAVrh74.MCK.GALGT2) will be delivered one time to each of the lower limbs through the femoral artery using an intravascular limb infusion technique (ILI)
Arm/Group | Cohort 1 (Minimal Efficacious Dose) rAAVrh74.MCK.GALGT2 | Cohort 1 rAAVrh74.MCK.GALGT2
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Minimal Efficacious Dose) rAAVrh74.MCK.GALGT2 (N=1) | Cohort 1 rAAVrh74.MCK.GALGT2 (N=1)
Bleeding at the femoral catheterization site (Vascular disorders) | 1 (1) | 0 (0) — Related to the Isolated Limb Infusion (ILI) procedure
Bruising (Vascular disorders) | 1 (1) | 1 (1) — Related to the Isolated Limb Infusion (ILI) procedure
Decrease in ejection fraction (Cardiac disorders) | 1 (1) | 0 (0) — Due to disease progression
Low Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Decreased Lymphocyte (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Cushingoid Face (Endocrine disorders) | 1 (1) | 0 (0) — Due to concomitant medication required by trial
Pharyngitis and Adenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Weight Gain (Endocrine disorders) | 1 (1) | 0 (0) — Due to concomitant medication required by trial
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) — Due to disease progression

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/90/NCT03333590/Prot_SAP_000.pdf